CLINICAL TRIAL: NCT03614156
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study of Rapastinel in the Prevention of Relapse in Patients With Major Depressive Disorder
Brief Title: Study of Monotherapy Rapastinel in the Prevention of Relapse in Patients With Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to stop the program.
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAP-MD-33; 2018-000064-28 (EudraCT Number)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorder, Major
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rapastinel weekly (Experimental): Rapastinel 450 mg or 225 mg (prefilled syringe, weekly intravenous IV administration)
  Interventions: Drug: Rapastinel
- Rapastinel clinically driven schedule (Experimental): Rapastinel 450 mg or 225 mg (prefilled syringe, clinically driven schedule IV administration, variable interval, placebo on intervening weeks)
  Interventions: Drug: Rapastinel
- Placebo weekly (Placebo Comparator): Placebo (prefilled syringe, weekly IV administration)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — Rapastinel 450 mg or 225 mg (prefilled syringe, weekly intravenous IV administration) or Rapastinel 450 mg or 225 mg (prefilled syringe, clinically driven schedule IV administration, variable interval, placebo on intervening weeks)
  Arms: Rapastinel clinically driven schedule; Rapastinel weekly
Drug: Placebo — Placebo (prefilled syringe, weekly IV administration)
  Arms: Placebo weekly

SUMMARY:
The study will evaluate the efficacy, safety, and tolerability of 450 milligrams (mg) or 225 mg of Rapastinel compared to placebo in the prevention of relapse in participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria: -

* Completion of Study RAP-MD-30, RAP-MD-31, or RAP-MD-32
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test

Exclusion Criteria: -

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1
* Lifetime history of meeting DSM-5 criteria for:
* 1.Schizophrenia spectrum or other psychotic disorder
* 2.Bipolar or related disorder
* 3.Major neurocognitive disorder
* 4.Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
* 5.Dissociative disorder
* 6.Posttraumatic stress disorder
* 7.MDD with psychotic features
* Significant suicide risk, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (52):
- United States (40):
  - Alea Research, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - California Pharmaceutical Research Institute, Anaheim, California
  - Synergy Research San Diego, National City, California
  - Excell Research Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Neuroscience Research Medical Group,Inc., Sherman Oaks, California
  - Viking Clinical Research Ltd., Temecula, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Research Centers of America, Hollywood, Florida
  - Clinical NeuroscienceSolutions, Inc., Jacksonville, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Innova Clinical Trials, Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Institute for Advanced Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Iris Research, Inc., Smyrna, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Pharmasite Research, Inc., Baltimore, Maryland
  - CBH Health, Gaithersburg, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Bioscience Research LLC, Mount Kisco, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Bugát Pál Hospital, Clinexpert, Gyöngyös, Hungary
- Japan (6):
  - Medical corporation Sato-Kai Yuge Hospital, Kumamoto
  - Sagaarashiyama-Tanaka Clinic, Kyoto
  - Sangenjaya Neurology- Psychosomatic Clinic, Setagaya-ku
  - Yoyogi Mental Clinic, Shibuya-ku
  - Maynds Tower Mental Clinic, Shibuya-ku
  - Ohwa Mental Clinic, Toshima-ku
- Centrum Medyczne Luxmed Sp.z o.o., Lublin, Poland
- Slovakia (4):
  - VAVRUŠOVÁ CONSULTING s.r.o., Psychiatrická ambulancia, Bratislava
  - MENTUM, s.r.o., Bratislava Mestská Časť Ružinov
  - Liptovská nemocnica s poliklinikou MUDr. Ivana Stodolu Liptovský Mikuláš, Liptovský Mikuláš
  - PsychoLine s.r.o., Psychiatrická ambulancia, Rimavská Sobota

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from RAP-MD-33 completed one of the rapastinel lead-in studies - RAP-MD-30, RAP-MD-31, or RAP-MD-32.
Pre-assignment Details: 363 patients enrolled in the Open Label Treatment Period (OLTP). Of these, 209 completed OLTP and 137 entered Double Blind Treatment Period (DBTP) and were randomized. Patients who completed or discontinued from the study can enter a 2-wk safety follow-up period (SFUP). 165 patients from OLTP and 91 patients from DBTP entered the SFUP.
Groups:
- Open-Label Treatment Period (OLTP) Weekly Rapastinel: Rapastinel 225 milligrams (mg) or 450 mg intravenous (IV) once a week during OLTP.
- DBTP Placebo Weekly: Placebo (prefilled syringe, weekly IV administration)
- DBTP Rapastinel Clinically Driven Schedule: Rapastinel 450 mg or 225 mg (prefilled syringe, clinically driven schedule IV administration, variable interval, placebo on intervening weeks)
- DBTP Rapastinel Weekly: Rapastinel 450 mg or 225 mg (prefilled syringe, weekly intravenous IV administration)
Period: Open-Label Treatment Period
Arm/Group | Open-Label Treatment Period (OLTP) Weekly Rapastinel | DBTP Placebo Weekly | DBTP Rapastinel Clinically Driven Schedule | DBTP Rapastinel Weekly
Started | 363 | 0 | 0 | 0
Completed | 209 | 0 | 0 | 0
Not Completed | 154 | 0 | 0 | 0
Not completed — Protocol-specified withdrawal met | 6 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0 | 0
Not completed — Lack of Efficacy | 18 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 36 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 74 | 0 | 0 | 0
Period: Double-Blind Treatment Period (DBTP)
Arm/Group | Open-Label Treatment Period (OLTP) Weekly Rapastinel | DBTP Placebo Weekly | DBTP Rapastinel Clinically Driven Schedule | DBTP Rapastinel Weekly
Started | 0 | 40 | 42 | 55
Completed | 0 | 10 | 11 | 10
Not Completed | 0 | 30 | 31 | 45
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 4
Not completed — Protocol Violation | 0 | 1 | 1 | 1
Not completed — Study terminated by sponsor | 0 | 22 | 26 | 38
Not completed — Miscellaneous Reasons | 0 | 1 | 0 | 0
Period: Safety Follow-Up Period
Arm/Group | Open-Label Treatment Period (OLTP) Weekly Rapastinel | DBTP Placebo Weekly | DBTP Rapastinel Clinically Driven Schedule | DBTP Rapastinel Weekly
Started | 165 | 26 | 30 | 35
Completed | 162 | 26 | 29 | 34
Not Completed | 3 | 0 | 1 | 1
Not completed — Miscellaneous Reasons | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Double-blind Safety Population consisted of all patients in the Open-label Safety Population who were randomized to a treatment group during the DBTP of the study and received at least 1 dose of double-blind IP.
Groups:
- Total: Total of all reporting groups
Arm/Group | DBTP Placebo Weekly | DBTP Rapastinel Clinically Driven Schedule | DBTP Rapastinel Weekly | Total
Number analyzed (Participants) | 40 | 42 | 55 | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47 (13.95) | 43.6 (12.57) | 43.9 (11.66) | 44.7 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 44 | 103
  Male | 10 | 13 | 11 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 9 | 20
  Not Hispanic or Latino | 37 | 34 | 46 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 8 | 5 | 11 | 24
  White | 27 | 33 | 42 | 102
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 84.84 (17.86) | 85.88 (19.21) | 88.53 (19.24) | 86.64 (18.77)
Height [Mean (Standard Deviation); unit: cm] | 168.31 (8.996) | 166.92 (9.858) | 168.47 (9.196) | 167.95 (9.304)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.89 (5.686) | 30.95 (7.289) | 31.15 (6.279) | 30.72 (6.421)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse During the 52 Weeks of the Double-Blind Treatment Period (DBTP)
Description: The time in days to first relapse is defined as the number of days from the date of randomization to the first relapse.
Time Frame: 52 Weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DBTP Placebo Weekly | DBTP Rapastinel Clinically Driven Schedule | DBTP Rapastinel Weekly
Number analyzed (Participants) | 40 | 42 | 55
Days | NA [NA to NA] — Not enough events to allow the estimation of the percentiles and the standard error for the confidence intervals. | 203 [177 to NA] — Not enough events to allow the estimation of the percentiles and the standard error for the confidence intervals. | NA [NA to NA] — Not enough events to allow the estimation of the percentiles and the standard error for the confidence intervals.

ADVERSE EVENTS:
Time Frame: The study consisted of an 8 to 16 week OLTP; followed by a randomized DBTP of up to 52 weeks; followed by a 2 week safety period.
Description: Adverse event data for non-randomized participants in the OLTP also include AEs that occurred during the safety follow period.
  Adverse event data for randomized participants in the DBTP were collected for up to 54 weeks which included the 2 week safety follow up period.
Groups:
- Open-Label Treatment Period: Rapastinel 225 milligrams (mg) or 450 mg intravenous (IV) once a week during OLTP.
Arm/Group | Open-Label Treatment Period | DBTP Placebo Weekly | DBTP Rapastinel Clinically Driven Schedule | DBTP Rapastinel Weekly
All-Cause Mortality (participants affected / at risk) | 0/363 | 0/40 | 0/42 | 0/55
Serious Adverse Events (participants affected / at risk) | 4/363 | 1/40 | 1/42 | 0/55
Other Adverse Events (participants affected / at risk) | 44/363 | 17/40 | 9/42 | 13/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Treatment Period (N=363) | DBTP Placebo Weekly (N=40) | DBTP Rapastinel Clinically Driven Schedule (N=42) | DBTP Rapastinel Weekly (N=55)
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Treatment Period (N=363) | DBTP Placebo Weekly (N=40) | DBTP Rapastinel Clinically Driven Schedule (N=42) | DBTP Rapastinel Weekly (N=55)
Nasopharyngitis (Infections and infestations) | 26 | 0 | 4 | 5
Headache (Nervous system disorders) | 20 | 3 | 1 | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 18 | 1 | 4 | 3
Nausea (Gastrointestinal disorders) | 4 | 2 | 1 | 2
Seasonal allergy (Immune system disorders) | 1 | 4 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 15 | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to study termination, the target number of participants needed to achieve target power and statistically reliable results was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03614156/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT03614156/SAP_001.pdf